CLINICAL TRIAL: NCT01231217
Title: Green Tea in Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GTCD-01
Record Dates: First submitted 2010-10-27; First posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Tea; Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- green (or white) tea (Other): Patients are recommended to drink green (or white) tea but are not allowed to consume any coffee
  Interventions: Other: Green tea (Camellia sinensis)
- coffee (Other): Patients are recommended to drink coffee but are not allowed to consume any tea
  Interventions: Other: Coffee

INTERVENTIONS:
Other: Green tea (Camellia sinensis) — Patients are recommended to drink at least 5 cups of green tea per day
  Arms: green (or white) tea
Other: Coffee — Patients are recommended to drink as much coffee as they tolerate.
  Arms: coffee

SUMMARY:
The purpose of this study is to assess whether green tea or coffee influence the course and life quality of patients with mild to moderately active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ≥ 18 years with signed informed consent,
* Patients with proven Crohn's disease,
* Chronic-active course ≥ 3 months,
* Current CDAI ≥ 150 and ≤ 350,
* All medications for Crohn's disease have to be on a constant dosage for at least 4 weeks prior to study entry (i.e. 5-ASA, steroids),
* Ability of the participant to understand character and individual consequences of the study.

Exclusion Criteria:

* Pregnancy or the wish to become pregnant, breastfeeding,
* Concomitant treatment with methotrexate, azathioprine or 6-mercaptopurine for < 3 months,
* Treatment with TNF-alpha-antagonists, cyclosporine or tacrolimus < 4 weeks prior to study entry,
* Participation in another study within the last 4 weeks,
* Ulcerative colitis or indeterminate colitis,
* Infectious colitis, including cytomegalovirus or Clostridium difficile induced colitis,
* Colitis for other reasons like known diverticulitis, radiation colitis, ischemic colitis or microscopic colitis,
* Malabsorption syndromes, lactose intolerance, celiac disease, exocrine pancreas insufficiency,
* Bleeding hemorrhoids,
* Other inflammatory or bleeding disorders of the colon and intestine, or diseases that may cause diarrhea or gastrointestinal bleeding,
* Intolerance / aversion to tea and/or coffee,
* Current treatment with antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-10

PRIMARY OUTCOMES:
Crohn's Disease Activity Index | week 16
  Assessment of clinical activity

SECONDARY OUTCOMES:
Harvey-Bradshaw-Index | week 16
  Assessment of clinical activity
Inflammatory Bowel Disease Questionnaire | week 16
  Assessment of Life Quality

CONTACTS AND LOCATIONS:
Overall Officials: Max Karner, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany